CLINICAL TRIAL: NCT05235321
Title: Automated Applanation Tonometry
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: device updates needed
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00106111
Record Dates: First submitted 2022-02-02; First posted 2022-02-11 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Glaucoma; Glaucoma, Suspect
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Intervention Model Description: In this study, 3 eye pressure measurements will be made in the upright position (standard GAT, fixed force GAT, upright applanating prototype) and 1 in the supine position (supine applanating prototype).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Standard GAT (Active Comparator): This is the standard method for IOP measurement in clinical practice
  Interventions: Device: Standard GAT
- Fixed-force GAT (Experimental): From the patient perspective, this method will feel identical to the standard GAT. The eye is given topical fluorescein/anesthetic. The GAT dial is set at 1.8 or 2.0, a C-MOS camera is connected to one of the oculars of the slit lamp machine and under blue light illumination, the GAT prism contacts the eye while the CMOS camera makes a video of the mire appearance through the ocular. The diameters of the recorded mire images are measured and the IOP is calculated based on the mire diameter
  Interventions: Device: Fixed force GAT
- Upright applanating prototype (Experimental): With this prototype, an applanating prism (custom manufactured with medical grade acrylic in an ISO-13485 certified facility) is attached to a fixed-force spring that creates a force equivalent to 1.8 or 2.0 on the GAT dial. Blue LED lights on the prototype are used to create the blue illumination similar to the blue light used in clinical practice on the slit lamp or Perkins tonometer. A C-MOS camera is aligned with the GAT prism to image the applanation mires. The eye is given topical fluorescein/anesthetic. Like fixed-force GAT, the GAT prism contacts the eye while the CMOS camera makes a video of the mire appearance. The diameters of the recorded mire images are measured and the IOP is calculated based on the mire diameter
  Interventions: Device: Upright applanating prototype
- Supine Applanating Prototype (Experimental): With this method, a 5 gram clear acrylic cylinder (custom manufactured with medical grade acrylic in an ISO-13485 certified facility) is aligned with the lens of the CMOS camera and the distal tip of the cylinder is illuminated with blue light using an LED similar to the blue light used in clinical practice on the slit lamp or Perkins tonometer. The eye is given topical fluorescein/anesthetic. While the CMOS camera is recording, the 5 gram weight will rest upon the eye and circular applanation mires are recorded. The diameters of the recorded mire images are measured and the IOP is calculated based on the mire diameter
  Interventions: Device: Supine Applanating Prototype

INTERVENTIONS:
Device: Standard GAT — Standard Goldmann Applanation Tonometry (GAT): this is the standard method for IOP measurement in clinical practice
  Arms: Standard GAT
Device: Fixed force GAT — An investigational device similar to standard GAT
  Arms: Fixed-force GAT
Device: Upright applanating prototype — An investigational device, prism used in standard and fixed-force GAT is attached to a portable device
  Arms: Upright applanating prototype
Device: Supine Applanating Prototype — An investigational device, prism used in standard and fixed-force GAT is attached to a portable device performed in the supine position
  Arms: Supine Applanating Prototype

SUMMARY:
Goldmann Applanation Tonometry (GAT) is considered the clinical gold standard for eye pressure measurements and yet it is known to be a subjective measurement with limited repeatability and limited portability. The purpose of this study is to develop an automated and objective method for performing applanation tonometry using standard ophthalmic equipment as well as using 2 portable prototypes.

DETAILED DESCRIPTION:
This is a prospective study. Patients presenting for their scheduled eye appointments will be recruited by verbal communication. Following informed consent, intraocular pressure (IOP) measurements will be made by the following 3 upright methods and 1 supine measurements:

1. Standard Goldmann Applanation Tonometry (GAT): this is the standard method for IOP measurement in clinical practice. The eye is given topical fluorescein/anesthetic, the GAT prism contacts the eye while the observer looks through the slit lamp machine ocular using blue light illumination to visual the applanation mires. The GAT dial is adjusted until mire alignment is achieved and the IOP measurement is read off the GAT dial.
2. Fixed force GAT: From the patient perspective, this method will feel identical to the standard GAT. The eye is given topical fluorescein/anesthetic. The GAT dial is set at 1.8 or 2.0, a complementary metal oxide semiconductor (C-MOS) camera is connected to one of the oculars of the slit lamp machine and under blue light illumination, the GAT prism contacts the eye while the CMOS camera makes a video of the mire appearance through the ocular. The diameters of the recorded mire images are measured and the IOP is calculated based on the mire diameter. A similar method using an iPod touch camera has been previously published by this PI.
3. Upright applanating prototype: With this prototype, an applanating prism (custom manufactured with medical grade acrylic in an ISO-13485 certified facility) is attached to a fixed-force spring that creates a force equivalent to 1.8 or 2.0 on the GAT dial. Blue LED lights on the prototype are used to create the blue illumination similar to the blue light used in clinical practice on the slit lamp or Perkins tonometer. A C-MOS camera is aligned with the GAT prism to image the applanation mires. The eye is given topical fluorescein/anesthetic. Like fixed-force GAT, the GAT prism contacts the eye while the CMOS camera makes a video of the mire appearance. The diameters of the recorded mire images are measured and the IOP is calculated based on the mire diameter.

   The order of the above 3 measurements will be randomized.

   The 4th measurement will be made with the patient in the supine position. Here, the subject will be reclined in our standard clinical exam chair until the iris plane is parallel to the ground.
4. Supine applanating prototype: With this method, a 5 gram clear acrylic cylinder (custom manufactured with medical grade acrylic in an ISO-13485 certified facility) is aligned with the lens of the CMOS camera and the distal tip of the cylinder is illuminated with blue light using an LED similar to the blue light used in clinical practice on the slit lamp or Perkins tonometer. The eye is given topical fluorescein/anesthetic. While the CMOS camera is recording, the 5 gram weight will rest upon the eye and circular applanation mires are recorded. The diameters of the recorded mire images are measured and the IOP is calculated based on the mire diameter. A similar method using an iPhone 6 camera has been previously published by this PI. The clear cylinder in this study is the same as that used in this prior study.

ELIGIBILITY:
Inclusion Criteria:

* Presenting for a routine eye exam
* ≥ 18 years of age
* Able and willing to give consent

Exclusion Criteria:

* History of corneal scarring
* Active infection of the eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure (IOP) as measured by standard GAT | Baseline
  this is the standard method for IOP measurement in clinical practice. The eye is given topical fluorescein/anesthetic, the GAT prism contacts the eye while the observer looks through the slit lamp machine ocular using blue light illumination to visual the applanation mires. The GAT dial is adjusted until mire alignment is achieved and the IOP measurement is read off the GAT dial.
Intraocular pressure (IOP) as measured by fixed force GAT | Baseline
  From the patient perspective, this method will feel identical to the standard GAT. The eye is given topical fluorescein/anesthetic. The GAT dial is set at 1.8 or 2.0, a C-MOS camera is connected to one of the oculars of the slit lamp machine and under blue light illumination, the GAT prism contacts the eye while the CMOS camera makes a video of the mire appearance through the ocular.
Intraocular pressure as measured by upright applanating | Baseline
  With this prototype, an applanating prism (custom manufactured with medical grade acrylic in an ISO-13485 certified facility) is attached to a fixed-force spring that creates a force equivalent to 1.8 or 2.0 on the GAT dial. Blue LED lights on the prototype are used to create the blue illumination similar to the blue light used in clinical practice on the slit lamp or Perkins tonometer. A C-MOS camera is aligned with the GAT prism to image the applanation mires. The eye is given topical fluorescein/anesthetic. Like fixed-force GAT, the GAT prism contacts the eye while the CMOS camera makes a video of the mire appearance. The diameters of the recorded mire images are measured and the IOP is calculated based on the mire diameter.
Intraocular pressure as measured by supine applanating protoype | Baseline
  With this method, a 5 gram clear acrylic cylinder (custom manufactured with medical grade acrylic in an ISO-13485 certified facility) is aligned with the lens of the CMOS camera and the distal tip of the cylinder is illuminated with blue light using an LED similar to the blue light used in clinical practice on the slit lamp or Perkins tonometer. The eye is given topical fluorescein/anesthetic. While the CMOS camera is recording, the 5 gram weight will rest upon the eye and circular applanation mires are recorded. The diameters of the recorded mire images are measured and the IOP is calculated based on the mire diameter.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Wen, MD, Principal Investigator — Duke Eye Center
Locations (1):
- Duke Eye Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No Currently, there is no plan to share data with other researchers.